CLINICAL TRIAL: NCT05443464
Title: A Phase I Safety Study of Single Dose Allogeneic Bone Marrow Derived MSCs for Steroid Refractory Acute Graft vs. Host Disease
Brief Title: Mesenchymal Stem Cells (MSCs) for Steroid Refractory Acute GVHD (SR-aGVHD)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: OSSM-001 will not be used in this program moving forward.
Sponsor: Ossium Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSSM-001-006-01
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: GVHD,Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 2M cells/kg (Experimental): Dose level 1. 3 subjects will receive OSSM-001 at 2M cells/kg and followed for 28 days post dose to observe for DLT.
  Interventions: Biological: OSSM-001
- 6M cells/kg (Experimental): Dose level 2. If no DLTs are observed in the previous dose level, 3 subjects will receive OSSM-001 at 6M cells/kg and followed for 28 days post dose to observe for DLT.
  Interventions: Biological: OSSM-001
- 12M cells/kg (Experimental): Dose level 3. If no DLTs are observed in the previous dose level, 3 subjects will receive OSSM-001 at 12M cells/kg and followed for 28 days post dose to observe for DLT.
  Interventions: Biological: OSSM-001
- 24M cells/kg (Experimental): Dose level 4. If no DLTs are observed in the previous dose level, 3 subjects will receive OSSM-001 at 24M cells/kg and followed for 28 days post dose to observe for DLT.
  Interventions: Biological: OSSM-001

INTERVENTIONS:
Biological: OSSM-001 — Direct IV infusion of OSSM-001

SUMMARY:
The objective of this clinical study is to demonstrate safety and feasibility of single-dose infusion of Ossium MSCs product (OSSM-001) to treat steroid refractory acute GVHD (SR-aGVHD).

DETAILED DESCRIPTION:
The dose escalation will be used to establish a maximum tolerated dose, starting from 2M cells/kg. If no safety issues are seen, then MSCs dose maybe escalated to 6M cells/kg, 12M cells/kg and 24M cell/kg based on data review from each cohort. Additional studies will be conducted to establish a dosing regimen and to evaluate the safety and efficacy of OSSM-001 for SR-aGVHD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum 18 years of age who have undergone hematopoietic cell transplantation (HCT), from any donor source donor (including HLA-matched related and unrelated, haploidentical and umbilical cord donors) with any conditioning regimen
2. Clinically diagnosed Grades II to IV acute GVHD as per standard criteria occurring within 100 days of HCT
3. Confirmed diagnosis of steroid refractory aGVHD defined as patients administered high-dose systemic corticosteroids (methylprednisolone 2 mg/kg/day [or equivalent prednisone dose 2.5 mg/kg/day]), given alone or combined with calcineurin inhibitors (CNI) and either:

   1. Progressing based on organ assessment after at least 3 days at the time of initiation of high-dose systemic corticosteroid +/- CNI for the treatment of Grade II-IV aGVHD, OR
   2. Failure to achieve at a minimum partial response based on organ assessment after 7 days compared to organ stage at the time of initiation of high-dose systemic corticosteroid +/- CNI for the treatment of Grade II-IV aGVHD, OR
   3. Patients who fail corticosteroid taper defined as fulfilling either one of the following criteria:

   i. Requirement for an increase in the corticosteroid dose to methylprednisolone ≥2 mg/kg/day (or equivalent prednisone dose ≥2.5 mg/kg/day), OR

   ii. Failure to taper the methylprednisolone dose to <0.5 mg/kg/day (or equivalent prednisone dose <0.6 mg/kg/day) for a minimum 7 days.
4. Minimum Karnofsky Performance Level of at least 30 or higher at the time of study entry.

Exclusion Criteria:

1. Has received more than one systemic treatment for steroid refractory aGVHD in addition to steroids.
2. Received stem cell therapy in the past
3. Presence of an active uncontrolled infection including significant bacterial, fungal, viral, or parasitic infection requiring treatment
4. Presence of relapsed primary malignancy, or who have been treated for relapse after the HCT was performed, or who may require rapid immune suppression withdrawal as pre-emergent treatment of early malignancy relapse.
5. Evidence of pulmonary infiltrate or hemorrhage based on imaging or requiring high flow oxygen via face mask
6. Patients who have had treatment with any other investigational agent, device, or procedure within 30days (or 5 half-lives, whichever is greater) prior to enrollment.
7. Patients who have received more than one HCT
8. Any medical or psychological condition or situation deemed by the Investigators to put the patient at increased risk of complications or non-compliance.
9. Unresolved veno-occlusive disease
10. HLA antibody screen positive for HLA antibodies specific against the MSCs products
11. ALT or AST > 5X of upper limit of normal
12. Serum Bilirubin >2 X of upper limit of normal
13. GFR <50 ml/min
14. SpO2 <94% despite being on continuous supplemental oxygen
15. Patients requiring continuous >4L/minute of supplemental oxygen (irrespective of oxygen saturation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-05 (Estimated); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-10-14 (Estimated)

PRIMARY OUTCOMES:
Safety events | 112 days (16 weeks)
  OSSM-001 related safety events

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) | 112 days (16 weeks)
  Determine MTD of OSSM-001

OTHER OUTCOMES:
Overall survival (OS) from initiation of therapy | 112 days (16 weeks)
  OS rate at day 112 post initiation of therapy
Overall survival (OS) by baseline GVHD grading | 112 days (16 weeks)
  OS rate at day 112 by baseline GVHD grading post initiation of therapy
Overall survival (OS) stratified by organ involvement | 112 days (16 weeks)
  OS rate at day 112 stratified by organ involvement post initiation of therapy
Overall disease relapse | 112 days (16 weeks)
  Overall disease relapse by day 112 post initiation of therapy
Overall opportunistic infection rate | 112 days (16 weeks)
  Overall opportunistic infection rate by day 112 post initiation of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Munjal, Study Director — Ossium Health, Inc.

IPD SHARING:
Plan to Share IPD: No